CLINICAL TRIAL: NCT05017545
Title: Measuring the Impact of Carfilzomib and Belatacept on Allogeneic Desensitization in Prospective Kidney Transplant Recipients (ITN089ST)
Brief Title: Carfilzomib and Belatacept for Desensitization
Acronym: ADAPT
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Immune Tolerance Network (ITN) (Network); Bristol-Myers Squibb (Industry); PPD Development, LP (Industry); Rho Federal Systems Division, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DAIT ITN089ST; ITN089ST (Other: Immune Tolerance Network (ITN)); NIAID CRMS ID#: 38685 (Other: DAIT NIAID)
Record Dates: First submitted 2021-08-17; First posted 2021-08-24 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Highly Sensitized Prospective Kidney Transplant Recipients
Keywords: calculated panel reactive antibodies (cPRA); desensitization therapy; human leukocyte antigen (HLA) desensitization
MeSH Terms: interventions — carfilzomib; Abatacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (N=5 Subjects) (Experimental): The two investigational agents used in this study are carfilzomib and belatacept.
  Per protocol, Carfilzomib administered intravenously:
  * Cycle 1 will consist of 2 doses in week 4 (Day 28 and 29). If tolerated, the dose will be increased and administered twice a week in weeks 5 (Day 35 and 36) and 6 (Day 42 and 43).
  * Cycle 2 will consist of a total of 6 doses, administered twice weekly in weeks 12 (Day 84 and 85), 13 (Day 91 and 92) and 14 (Day 98 and 99).
  Per protocol, Belatacept:
  -Belatacept will be administered intravenously on days 29 (week 4), 33 (week 5), and weeks 6, 8, 12, 16, then at a lower dose at week 20, 24, 28, 32, 36, 40, 44, 48, 52, and 56. Dosing is based on the recommended dose in the package insert.
  Interventions: Biological: carfilzomib; Biological: belatacept; Procedure: Bone marrow aspiration
- Cohort 2 (N=10 Subjects) (Experimental): The enrollment of ten additional subjects and dosing regimen is dependent on the results in Cohort 1.°
  Per protocol, Carfilzomib administered intravenously:
  * Cycle 1 will consist of 2 doses in week 4 (Day 28 and 29). If tolerated, the dose will be increased and administered twice a week in weeks 5 (Day 35 and 36) and 6 (Day 42 and 43).
  * Cycle 2 will consist of a total of 6 doses, administered twice weekly in weeks 12 (Day 84 and 85), 13 (Day 91 and 92) and 14 (Day 98 and 99).
  Per protocol, Belatacept:
  -Belatacept will be administered intravenously on days 28 (week 4), 33 (week 5), and weeks 6, 8, 12, 16, then at a lower dose at week 20, 24, 28, 32, 36, 40, 44, 48, 52, and 56. Dosing is based on the recommended dose in the package insert.
  ° May be modified based on the safety and efficacy analysis of Cohort 1.
  Interventions: Biological: carfilzomib; Biological: belatacept; Procedure: Bone marrow aspiration

INTERVENTIONS:
Biological: carfilzomib — Administered: Intravenously (IV). Carfilzomib is administered intravenously, on two consecutive days, each week for three weeks per cycle. In this study, subjects will receive 2 cycles of carfilzomib. Dosing for each cycle is based on the recommended dosing for carfilzomib monotherapy in the package insert.
  Carfilzomib is a proteasome inhibitor indicated for the treatment of patients with multiple myeloma. In this study, carfilzomib will be used in highly sensitized subjects without myeloma who are awaiting a kidney transplant.
  Other Names: Kyprolis®
Biological: belatacept — Administered: Intravenously (IV). Belatacept is indicated for the prophylaxis of organ rejection in adult patients receiving a kidney transplant. In this study, belatacept will be used in highly sensitized subjects who are awaiting a kidney transplant.
  Other Names: Nulojix®
Procedure: Bone marrow aspiration — Subjects will undergo a bone marrow aspiration prior to starting the study regimen and at 16 weeks after starting the study regimen. In subjects who undergo a kidney transplant during the study, another bone marrow aspiration will be done if it has been >4 weeks since the previous bone marrow aspiration.

SUMMARY:
Some kidney transplant candidates have a very low chance of getting a kidney transplant because their immune systems are "highly sensitized" to most kidney donors. Being "highly sensitized" means that they will likely have to wait a long time (more than 5 years) before an acceptable donor is found for them or, they never receive a compatible donor, and die while on the kidney transplant waitlist.

The purpose of this study is to find out whether two drugs, carfilzomib (Kyprolis®),and belatacept (Nulojix®), can make these kidney transplant candidates less sensitized, and make it easier and quicker to find a kidney donor for them.

DETAILED DESCRIPTION:
This study will enroll 15 eligible participants, 18 to 65 years of age, with end stage renal failure on dialysis who are on the waiting list for a deceased donor transplant with calculated panel reactive antibodies (cPRA) ≥99.9% or >98% (with >5 years of waiting time) or, those with cPRA >98% and an human leukocyte antigen (HLA)-incompatible approved living donor who have not received a transplant after 1 year in a paired kidney exchange program. The study will evaluate whether the study treatment is safe and can lower the participant's immune system's sensitization to kidney donors, making it easier to find a well-matched kidney for them.

Participants in the study will be enrolled in two consecutive Cohorts of 5 and 10 patients respectively. The total duration of participation in the study will be 76 weeks for Cohort 1 and 68 weeks for Cohort 2. Participants who undergo kidney transplantation while enrolled in the study will have 52 weeks of follow up post-transplant.

The duration of participation for living donors is one study visit. Their participation in the study ends upon completion of this study visit.

ELIGIBILITY:
Inclusion Criteria:

Individuals who meet all of the following criteria are eligible for enrollment as study subjects-

1. Subject must be able to understand and provide informed consent
2. End stage renal disease (ESRD) on dialysis
3. United Network for Organ Sharing (UNOS) listed for a kidney transplant with any one of the following:

   * Current calculated panel reactive antibodies (cPRA) ≥ 99.9 percent awaiting deceased donor transplant
   * Current cPRA >98 percent (with >5 years of waiting time) awaiting deceased donor transplant
   * Current cPRA >98 percent with Human Leukocyte Antigen (HLA)-incompatible approved living donor and has not received a transplant after 1 year in a kidney paired exchange program
4. Evidence of established immunity to Epstein-Barr virus (EBV) as demonstrated by serologic testing
5. Negative result of most recent tuberculosis (TB) testing or appropriately completed latent tuberculosis infection (LTBI) therapy.

   * Testing should be conducted using either a purified protein derivative (PPD) or interferon-gamma release assay (i.e. QuantiFERON-TB, T-SPOT.TB).
   * Negative results from tests performed within 12 months prior to study entry are acceptable in the absence of any intervening exposure to TB.
   * Subjects with a positive test result must have completed appropriate therapy for LTBI.

     * Note: LTBI treatment regimens should be among those endorsed by the Centers for Disease Control and Prevention (CDC), url: https://www.cdc.gov/tb/topic/treatment/ltbi.htm
6. Negative Food and Drug Administration (FDA)-approved test for human immunodeficiency virus (HIV) diagnosis (at screening or as documented in medical record, up to 6 months prior to screening)
7. Negative Hepatitis C antibody test at screening or as documented in medical record, up to 6 months prior to screening.

   --If there is a history of treated hepatitis C then documentation of two consecutive negative HCV quantitative ribonucleic acid (RNA) polymerase chain reaction (PCR) tests separated by at least 6 months is required. Untreated subjects with positive HCV antibody and a single negative HCV quantitative HCV RNA are eligible.
8. Negative result for SARS-CoV-2 by an FDA-authorized molecular diagnostic test. Examples include, but are not limited to RT-PCR, LAMP, TMA, and qSTAR.
9. Subjects must have an echocardiogram within the previous 1 year without any of the following findings:

   * severe left ventricular hypertrophy (LVH)
   * greater than mild LVH accompanied by diastolic dysfunction
   * left ventricular ejection fraction <40 percent
   * pulmonary hypertension defined as right ventricular systolic pressure >35 mm Hg or tricuspid regurgitant velocity >2.8 m/s
10. Female subjects of reproductive potential must have a negative pregnancy test upon study entry
11. All subjects of reproductive potential must agree to use contraception for the duration of the study
12. Subjects must have current vaccinations or documented immunity to:

    * varicella (chickenpox)
    * measles
    * hepatitis B
    * pneumococcus
    * influenza, and
    * varicella zoster (if ≥ 50 years old).

      * Note: If subjects require administration of either live or killed vaccines to meet eligibility requirements, they must wait at least 2 weeks between vaccination and the baseline visit (i.e., at least 4 weeks before initiation of therapy)

Living Donor Inclusion Criteria:

Living donors must meet all of the following criteria to be eligible-

1. Able to understand and provide informed consent for research
2. Meets United Network for Organ Sharing (UNOS) requirements for kidney organ donation

Exclusion Criteria:

Individuals who meet any of these criteria are not eligible for enrollment as study subjects-

1. Inability or unwillingness of a subject to give written informed consent or comply with study protocol
2. Known active current or history of invasive fungal infection, non-tuberculous mycobacterial infection
3. Hepatitis B surface antigen or core antibody positive
4. Serious uncontrolled concomitant major organ disease, excluding kidney failure
5. Chronic respiratory failure
6. Uncontrolled systemic hypertension
7. Previous non-kidney solid organ transplant or bone marrow transplant
8. Any infection requiring hospitalization and intravenous (IV) therapy within 4 weeks of screening or oral therapy within 2 weeks of screening
9. Primary or secondary immunodeficiency
10. History of thromboembolism (except thrombosis of dialysis vascular access site)
11. Subjects with myocardial infarction within 12 months of screening or cardiac dysrhythmias uncontrolled by medications
12. History of plasma cell dyscrasia
13. Known bleeding diathesis or coagulation abnormality
14. History of active tuberculosis (TB) (even if treated)
15. Malignancy within the last 5 years except treated basal and squamous cell cancer of the skin or treated cervical cancer in situ
16. Women who are currently pregnant or nursing
17. Alcohol, drug, or chemical abuse within 1 year
18. Treatment with any investigational agent within 4 weeks (or 5 half-lives of investigational drug, whichever is longer) of screening
19. Current treatment with other biological drug. If the potential subject receives standard of care antibody treatments for prophylaxis of COVID-19 (permitted in protocol), there must be a minimum interval of 2 weeks after this treatment and before initiation of the study therapy.
20. Current treatment with any medication which increases the risk of thromboembolic events including oral contraceptives
21. Currently smoking tobacco
22. Neutropenia (absolute neutrophil count <1000/microliter) or thrombocytopenia (platelet count <100,000/microliter) within 4 weeks prior to screening
23. Alanine Aminotransferase (ALT) or aspartate aminotransferase (AST) ≥3 times upper limit of normal (ULN) or total bilirubin ≥ 2 times ULN
24. Past or current medical problems or findings from physical examination or laboratory testing not listed above, which, in the opinion of the investigator, may:

    * pose additional risks from participation in the study
    * interfere with the subject's ability to comply with study requirements, or
    * impact the quality or interpretation of the data obtained from the study.

Exclusion Criteria for Living Donors:

1. There are no exclusion criteria for living donors.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-12-28 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects who do not meet a stopping rule for safety and remain free of all safety events listed in the outcome description, through Week 20 (Cohort 1) post treatment initiation or until receiving a transplant, whichever occurs earlier. | Up to 20 weeks post treatment initiation
  Proportion of subjects who have not met a subject stopping rule, and remain free of all of the following through Week 20 post treatment initiation or until receiving a transplant, whichever occurs earlier:
  1. Grade 3 or higher infusion reaction,
  2. Grade 3 or higher infections, and
  3. Any malignancy.
  The study site will grade the severity of adverse events experienced by the study subjects according to the criteria set forth in the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 (Published November 27, 2017).
Proportion of subjects who do not meet a stopping rule for safety and remain free of all safety events listed in the outcome description, through Week 24 (Cohort 2) post treatment initiation or until receiving a transplant, whichever occurs earlier. | Up to 24 weeks post treatment initiation
  Proportion of subjects who have not met a subject stopping rule, and remain free of all of the following through Week 24 post treatment initiation or until receiving a transplant, whichever occurs earlier:
  1. Grade 3 or higher infusion reaction,
  2. Grade 3 or higher infections, and
  3. Any malignancy.
  The study site will grade the severity of adverse events experienced by the study subjects according to the criteria set forth in the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 (Published November 27, 2017).
Proportion of subjects who meet any one of the pre-specified events detailed in the outcome description: from Baseline to Week 20 post treatment initiation - Cohort 1 | Baseline (Visit 0) to Week 20 post treatment initiation
  Proportion of subjects who meet any one of the following compared to Baseline (Visit 0):
  1. Elimination of one human leukocyte antigen (HLA) antibody at Week 20 (which is Study Week 24) post treatment initiation,
  2. 50% or greater reduction in the mean fluorescence intensity (MFI) of at least three HLA antibodies at Week 20 (which is Study Week 24) after starting treatment, and/or
  3. Kidney transplant with a previously incompatible donor within 20 weeks after starting treatment without graft loss due to acute antibody mediated rejection occurring within the first four weeks post-transplant and caused by an anamnestic response.
Proportion of subjects who meet any one of the pre-specified events detailed in the outcome description: from Baseline to Week 24 post treatment initiation - Cohort 2 | Baseline (Visit 0) to Week 24 post treatment initiation
  Proportion of subjects who meet any one of the following compared to Baseline (Visit 0):
  1. Elimination of one human leukocyte antigen (HLA) antibody at Week 24 (which is Study Week 28) post treatment initiation,
  2. 50% or greater reduction in the mean fluorescence intensity (MFI) of at least three HLA antibodies at Week 24 (which is Study Week 28) after starting treatment, and/or
  3. Kidney transplant with a previously incompatible donor within 52 weeks after starting treatment without graft loss due to acute antibody mediated rejection occurring within the first four weeks post-transplant and caused by an anamnestic response.

SECONDARY OUTCOMES:
Proportion of subjects transplanted with a previously incompatible donor within 52 weeks after starting treatment | Within 52 weeks post treatment initiation
  Clinical outcome measure.
  Subjects may receive a kidney transplant while in the study, either from a living or deceased donor to whom they were previously compatible, or from a previously incompatible donor in case there is a significant reduction in HLA antibody.
Proportion of subjects with biopsy-proven acute or chronic antibody mediated rejection (AMR) within 52 weeks post-transplant in subjects who undergo a kidney transplant | Within 52 weeks post-transplant
  Clinical outcome measure.
  Antibody mediated rejection (AMR) is an important cause of graft loss after organ transplantation and is caused by anti-donor-specific antibodies, especially anti- human leukocyte antigen (HLA) antibodies.
Number of biopsy-proven acute or chronic AMR events within 52 weeks post-transplant in subjects who undergo a kidney transplant | Within 52 weeks post-transplant
  Clinical outcome measure.
  Antibody mediated rejection (AMR) is an important cause of graft loss after organ transplantation and is caused by anti-donor-specific antibodies, especially anti- human leukocyte antigen (HLA) antibodies.
Incidence of invasive fungal infections, mycobacterial infections or Pneumocystis jirovecii infection within 20 weeks after starting treatment - Cohort 1 | Within 20 weeks post treatment initiation
  A measure of infection-related morbidity.
Incidence of invasive fungal infections, mycobacterial infections or Pneumocystis jirovecii infection within 24 weeks after starting treatment - Cohort 2 | Within 24 weeks post treatment initiation
  A measure of infection-related morbidity.
Incidence of invasive fungal infections, mycobacterial infections or Pneumocystis jirovecii infection within 52 weeks after starting treatment | Within 52 weeks post treatment initiation
  A measure of infection-related morbidity.
Incidence of cytomegalovirus (CMV) infection within 20 weeks after starting treatment (Cohort 1) | Within 20 weeks post treatment initiation
  CMV infection confirmed by the presence of detectable CMV in blood by polymerase chain reaction [PCR] diagnostic testing, regardless of whether signs or symptoms are present.
Incidence of cytomegalovirus (CMV) infection within 24 weeks after starting treatment (Cohort 2) | Within 24 weeks post treatment initiation
  CMV infection confirmed by the presence of detectable CMV in blood by polymerase chain reaction [PCR] diagnostic testing, regardless of whether signs or symptoms are present.
Incidence of cytomegalovirus (CMV) infection within 52 weeks after starting treatment | Within 52 weeks post treatment initiation
  CMV infection confirmed by the presence of detectable CMV in blood by polymerase chain reaction [PCR] diagnostic testing, regardless of whether signs or symptoms are present.
Incidence of cytomegalovirus (CMV) disease within 20 weeks after starting treatment | Within 20 weeks post treatment initiation
  CMV disease defined by the presence of detectable CMV in the blood and the presence of other clinical manifestations attributable to the CMV virus.
Incidence of cytomegalovirus (CMV) disease within 52 weeks after starting treatment | Within 52 weeks post treatment initiation
  CMV disease defined by the presence of detectable CMV in the blood and the presence of other clinical manifestations attributable to the CMV virus.
Incidence of post-transplant lymphoproliferative disorder (PTLD) | Within 52 weeks post-transplant
  As per diagnosis by local pathologist and treating physician.
Mean number of Human Leukocyte Antigen (HLA) antibodies eliminated, compared to Baseline (Cohort 1) | Baseline (Visit 0), Weeks 16, 20, and 52 post treatment initiation
  Mechanistic outcome measure focusing on change in donor specific antibodies (DSA).
Mean number of Human Leukocyte Antigen (HLA) antibodies eliminated, compared to Baseline (Cohort 2) | Baseline (Visit 0), Weeks 16, 24, and 52 post treatment initiation
  Mechanistic outcome measure focusing on change in donor specific antibodies (DSA).
Mean proportion of Human Leukocyte Antigen (HLA) antibodies eliminated, compared to Baseline (Cohort 1) | Baseline (Visit 0), Weeks 16, 20, and 52 post treatment initiation
  Mechanistic outcome measure focusing on change in donor specific antibodies (DSA).
Mean proportion of Human Leukocyte Antigen (HLA) antibodies eliminated, compared to Baseline (Cohort 2) | Baseline (Visit 0), Weeks 16, 24, and 52 post treatment initiation
  Mechanistic outcome measure focusing on change in donor specific antibodies (DSA).
Mean percent reduction from Baseline in mean fluorescence intensity (MFI) of the immunodominant Human Leukocyte Antigen (HLA) antibody, Class I and Class II - only collected for Cohort 1 | Baseline (Visit 0), Weeks 16, 20, and 52 post treatment initiation
  Mechanistic outcome measure focusing on change in donor specific antibodies (DSA).
Mean percent reduction from Baseline in mean fluorescence intensity (MFI) of Human Leukocyte Antigen (HLA) antibodies classified by an MFI >10,000 at treatment initiation (Cohort 1) | Baseline (Visit 0), Weeks 16, 20, and 52 post treatment initiation
  Mechanistic outcome measure focusing on change in donor specific antibodies. An MFI of >10,000 reflects a strong DSA intensity. (Reference: A measure of 0 reflects no donor specific antibodies).
Mean percent reduction from Baseline in mean fluorescence intensity (MFI) of Human Leukocyte Antigen (HLA) antibodies classified by an MFI >10,000 at treatment initiation (Cohort 2) | Baseline (Visit 0), Weeks 16, 24, and 52 post treatment initiation
  Mechanistic outcome measure focusing on change in donor specific antibodies. An MFI of >10,000 reflects a strong DSA intensity. (Reference: A measure of 0 reflects no donor specific antibodies).

CONTACTS AND LOCATIONS:
Overall Officials: Stuart J. Knechtle, MD, Study Chair — Duke Department of Surgery, Duke University School of Medicine; Annette M. Jackson, PhD, Study Chair — Duke Department of Surgery, Duke University School of Medicine
Locations (1):
- Duke Transplant Center, Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
The plan is to share data upon completion of the study in: Immunology Database and Analysis Portal (ImmPort), a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts.
Time Frame: On average, within 24 months after database lock for the trial.
Access Criteria: Open access.
URL: https://www.immport.org/home

REFERENCES:
- See also: Immune Tolerance Network — https://www.immunetolerance.org/
- See also: National Institute of Allergy and Infectious Diseases — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation — https://www.niaid.nih.gov/about/dait